CLINICAL TRIAL: NCT02787330
Title: Assessing the Efficacy of a Psychosocial Intervention Program for Siblings of Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Maru Barrera, Psychologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000028990
Record Dates: First submitted 2016-05-09; First posted 2016-06-01 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Cancer
Keywords: pediatric cancer; psychosocial; siblings
MeSH Terms: conditions — Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): Behavioural: Participants in this arm will experience an 8-week manualized intervention program with activities and games. Sessions will NOT be designed around a specific theme related to childhood cancer and sibling relationships. Activities and games will NOT have a specific focus. Sessions will be conducted by facilitators who will receive the standard training for volunteers and will work under the supervision of one of the investigators at each site.
  Interventions: Behavioral: Control Group
- Experimental Group (Experimental): Behavioural: Participants in this arm will experience an 8-week manualized intervention program which focuses on education, therapeutic problem solving, and social support. Each intervention session is structured by theme relevant to the cancer experience and themes are addressed through fun activities, games, arts, and crafts.To maximize the therapeutic effect of the intervention fun work (homework) will be assigned after each session. Training for the EG facilitators requires reading and studying the manual to become fully familiarized with the intervention approaches, observing group sessions through a one-way mirror prior to participation as a group facilitator, and participating as a group facilitator assistant for the intervention program.
  Interventions: Behavioral: Experimental Group

INTERVENTIONS:
Behavioral: Control Group — Sessions will not be designed around a specific theme related to childhood cancer and sibling relationships. Activities and games will not have a specific focus. CG sessions will be conducted by facilitators who will receive the standard training for volunteers and will work under the supervision of one of the investigators at each site.
  Arms: Control Group
Behavioral: Experimental Group — The experimental group will be detailed, session by session, in the manual written for this purpose. It addresses on topic per session (respecting each other, medical information about cancer, family relationships, sibling's fears and feelings, relationship between siblings, relationships at school, generating hope.
  Arms: Experimental Group

SUMMARY:
The psychosocial effects of childhood cancer and its demanding medical treatment can affect not only the ill child but the whole family, particularly siblings who are often overlooked given the terrible circumstances these families face. Current evidence suggests that negative long-term psychosocial effects of childhood cancer may be more severe in siblings than in the child with cancer. Addressing these effects on siblings may benefit the child with cancer and the entire family. Thus, early psychosocial preventive interventions are needed to foster psychosocial adjustment in siblings and promote better quality of life for the entire family. The immediate objective of this study is to address siblings' psychological distress by assessing feasibility and efficacy of a manualized group intervention for siblings of children with cancer (Siblings Coping Together, SibCT). A longer term objective is that the evidence-based intervention could then be exported to other centres across Canada and internationally. Additionally, the study results will identify biomedical, personal, familial and social determinants of intervention outcomes that can guide clinical effort for those at greatest risk. Finally, the overall aim of the project is to reduce psychological distress and improve quality of life for siblings and families impacted by a cancer diagnosis and its demanding treatment.

DETAILED DESCRIPTION:
Siblings of children with cancer can endure great psychological distress as a result of their brother's or sister's diagnosis and treatment. Understandably, when a child has cancer, their parents' attention is focused mainly on that child and therefore the siblings' needs may not be fully addressed. Thus, siblings often develop feelings of anger, abandonment, jealousy, and fear, which may lead to an increased risk for academic difficulties, symptoms of depression and anxiety and post traumatic stress disorder, although the results are not consistent across studies. Of most concern is that psychological problems may persist through adulthood, as suggested by a recent study in which alcoholism was more prevalent among siblings of children with cancer when compared to peers and cancer survivors. Therefore, it is imperative to develop evidence based psychological intervention programs to prevent these detrimental psychological effects in siblings of children with cancer. This project aims to address siblings' psychological distress by assessing the efficacy of a manualized group intervention for siblings of children with cancer (SibCT) across three Canadian sites (SickKids, Alberta Children's Hospital, BC Women and Children's Hospital) using a randomized control trial (RCT) experimental design. A manualized intervention is considered the gold standard for psychological intervention as it ensures replicability of the study and intervention fidelity. The primary aim is to demonstrate that survivors in the SibCT group (EG) demonstrate decreased symptoms of depression and anxiety improve their overall quality of life compared to an attention control group (CG). A secondary aim is to show that compared to CG, EG will show improvements in secondary measures of quality of life as well as knowledge about cancer. We will also explore other factors such as disease and treatment variables, social contextual variables, individual (sibling) variables and family variables. Randomized Control Trial design with repeated measures will be used. Siblings of children on active cancer treatment and at least 3 months from diagnosis to reduce parental burden; between 8-16 years of age will be included in the study. Siblings will be randomized to either the EG or CG. Approximately 184 siblings will be recruited across the three pediatric centres. After baseline assessment, both groups will have 8 two-hour weekly group sessions consisting of arts and crafts and games, and two post-intervention assessments; at the end of session 8 and three months later. In the EG the critical ingredient has education and social and therapeutic problem solving components based on the manual. Examples of weekly session topics include: age-appropriate medical information about cancer; siblings' fears and feelings; relationships at school, etc. The CG will not have any education or therapeutic-based components. Rigorous testing of the efficacy of an intervention program is a critical step for developing evidence-based treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Siblings of children on active cancer treatment at one or the three sites; at least three months from diagnosis to reduce parental burden
2. Siblings and one caregiver are fluent in English, ensuring full participation
3. Siblings are age 8-16 years

Exclusion Criteria:

1. Siblings who are diagnosed with a developmental or psychiatric disorder which will prevent full group participation
2. Are receiving active psychological treatment at the time of recruitment
3. Has a brother/sister who is receiving palliative care, and is not expected to live longer than 6 months or who had died.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline depression scores at end of intervention and 3 months | day 1, 8 weeks later, and 3 months after day 1
  Measured by Childhood Depression Inventory (CDI) [Kovacs, 1992]. ). This self-rated, 27-item scale was designed for children between the ages of 7-17.
Change from baseline anxiety scores at end of intervention and 3 months | day 1, 8 weeks later, and 3 months after day 1
  Measured by State Trait Anxiety Inventory for Children (STAIC)( Spielberger, 1983). This is a 20-item self-report measure

SECONDARY OUTCOMES:
knowledge about cancer | day 1, 8 weeks later, and 3 months after day 1
  Siblings Perception Questionnaire (SPQ) (Barbarin, 1995) is a 17-item questionnaire specifically designed for siblings of children with cancer
quality of life | day 1, 8 weeks later, and 3 months after day 1
  Pediatric Quality of Life Inventory (PedsQL 4.0 Varni, 1999) is a 23-item, standardized generic measure of health related QOL. The PedsQL, self-report and parent proxy, is composed of four subscales: Physical, Social, Emotional and School Functioning and a Total score.

OTHER OUTCOMES:
exploratory outcome, maternal distress | day 1, 8 weeks later, and 3 months after day 1
  Multidimensional Anxiety Questionnaire, (MAQ) (Reynolds, 1999). MAQ consists of 40 items.
perceived social support | day 1, 8 weeks later, and 3 months after day 1
  Perceived social support will be assessed as a potential social determinant of siblings' outcomes, using the Social Support Scale for Children (SSSC) (Harter, 1985). This scale has 24 items assessing 8 to 17-year-old children's perceptions of social support from others, including parents, teachers, classmates, and close friends.

CONTACTS AND LOCATIONS:
Overall Officials: Maru Barrera, PhD, Principal Investigator — The Hospital for Sick Children
Locations (3):
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Women and Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrera, M, Chung, JJ, Greenberg, M & Fleming, CF. Preliminary investigation of a group intervention for siblings of pediatric cancer patients. Children's Health Care, 31(2), 131-142, 2002.
- [Background] Alderfer MA, Labay LE, Kazak AE. Brief report: does posttraumatic stress apply to siblings of childhood cancer survivors? J Pediatr Psychol. 2003 Jun;28(4):281-6. doi: 10.1093/jpepsy/jsg016. PMID 12730285
- [Background] Alderfer MA, Hodges JA. Supporting Siblings of Children with Cancer: A Need for Family-School Partnerships. School Ment Health. 2010 Jun 1;2(2):72-81. doi: 10.1007/s12310-010-9027-4. PMID 20582154
- [Background] Barrera, M., Chung, J. J., & Fleming, C. F. (2004). A group intervention for siblings of pediatric cancer patients. Journal of Psychological Oncology, 22(2), 21-39.
- [Background] Sidhu R, Passmore A, Baker D. The effectiveness of a peer support camp for siblings of children with cancer. Pediatr Blood Cancer. 2006 Oct 15;47(5):580-8. doi: 10.1002/pbc.20653. PMID 16317733
- [Background] Kamibeppu K, Sato I, Honda M, Ozono S, Sakamoto N, Iwai T, Okamura J, Asami K, Maeda N, Inada H, Kakee N, Horibe K, Ishida Y. Mental health among young adult survivors of childhood cancer and their siblings including posttraumatic growth. J Cancer Surviv. 2010 Dec;4(4):303-12. doi: 10.1007/s11764-010-0124-z. Epub 2010 Apr 16. PMID 20396974
- [Background] Packman W, Weber S, Wallace J, Bugescu N. Psychological effects of hematopoietic SCT on pediatric patients, siblings and parents: a review. Bone Marrow Transplant. 2010 Jul;45(7):1134-46. doi: 10.1038/bmt.2010.74. Epub 2010 Apr 12. PMID 20383219
- [Background] Lown EA, Goldsby R, Mertens AC, Greenfield T, Bond J, Whitton J, Korcha R, Robison LL, Zeltzer LK. Alcohol consumption patterns and risk factors among childhood cancer survivors compared to siblings and general population peers. Addiction. 2008 Jul;103(7):1139-48. doi: 10.1111/j.1360-0443.2008.02242.x. PMID 18554347